CLINICAL TRIAL: NCT00827268
Title: Multimodal Treatment of Phonological Alexia: Behavioral & fMRI Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B6699-W
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Aphasia; Stroke; Dyslexia, Acquired
Keywords: Dyslexia; Reading; Aphasia; Stroke
MeSH Terms: conditions — Aphasia; Stroke; Dyslexia, Acquired; Dyslexia

STUDY DESIGN:
Intervention Model Description: This is a repeated probe design study.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other): Repeated probes every 8 hours of treatment (1/week)
  Interventions: Behavioral: One-on-one treatment of reading difficulties

INTERVENTIONS:
Behavioral: One-on-one treatment of reading difficulties — Multimodal behavioral treatment focused on retraining sound to letter associations and skills in sounding out words when reading. Treatment has been pilot-tested in published papers since 1998.

SUMMARY:
This study offers 90-120 hours of 1:1 training to improve reading skills in adults who have poor reading skills following a stroke. Specifically, this study is designed to improve skill in sounding out words for reading and spelling. The overall time commitment for participation in this study is approximately 11-30 weeks.

DETAILED DESCRIPTION:
The proposed study is a mixed-effects (single-subject ABA repeated-probe and small group elements) design with 90-120 hours of a modified multi-modal treatment of alexia replicated across up to 18 adults with post-stroke phonological alexia. The short-term goals of this research proposal includes the following: 1) determine if a modified multimodal treatment of phonological alexia can improve pseudoword reading skills (providing a basis from which training will also treat real word reading skills), 2) determine if a modified multimodal treatment of phonological alexia can improve real word reading skills, 3) determine how brain lesion extent and location relate to participants' response to treatment, and 4) identify relationships between changes in functional brain activity in specified regions of interest and participants' response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults with post-stroke reading difficulties (phonological alexia)
* >3 months post-stroke
* native English speaker
* can go in MRI scanner (3 to 6 scans),
* participate in 90 to 120 free treatment sessions
* return for 3-month post-treatment follow-up assessment & MRI.

Exclusion Criteria:

* mental illness
* degenerative disease, visual or auditory acuity impairment
* drug abuse
* English is not first language
* claustrophobia
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in Real World Reading Skills | Language testing are conducted two weeks prior to treatment, immediately following end of treatment and 3 months after end of treatment.
  Real World Reading Skills was tested using the Woodcock Reading Mastery Test-Revised

CONTACTS AND LOCATIONS:
Overall Officials: Timothy W. Conway, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States

REFERENCES:
- See also: Dr. Conway's homepage — http://neuropsy.phhp.ufl.edu/facres/facprofiles/Conway.html